CLINICAL TRIAL: NCT02037295
Title: Investigation of the Gut Microbiota in Regulating Nutrient Absorption in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 999914045; 14-DK-N045 (Other: NIDDK)
Record Dates: First submitted 2014-01-14; First posted 2014-01-15 (Estimated); Results first posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2019-03-29

CONDITIONS: Obesity
Keywords: Gut Microbiota; Obesity; Absorption; Overfeeding
MeSH Terms: conditions — Obesity | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- OF_UF Vancomycin (Experimental): Healthy volunteers assigned overfeeding diet, underfeeding diet, and then vancomycin
  Interventions: Drug: Vancomycin; Other: Overfeeding diet (OF); Other: Underfeeding diet (UF)
- OF_UF Placebo (Placebo Comparator): Healthy volunteers assigned overfeeding diet, underfeeding diet, and then placebo
  Interventions: Drug: Placebo oral tablet; Other: Overfeeding diet (OF); Other: Underfeeding diet (UF)
- UF_OF Vancomycin (Experimental): Healthy volunteers assigned underfeeding diet, overfeeding diet, and then vancomycin
  Interventions: Drug: Vancomycin; Other: Overfeeding diet (OF); Other: Underfeeding diet (UF)
- UF_OF Placebo (Placebo Comparator): Healthy volunteers assigned underfeeding diet, overfeeding diet, and then placebo
  Interventions: Drug: Placebo oral tablet; Other: Overfeeding diet (OF); Other: Underfeeding diet (UF)

INTERVENTIONS:
Drug: Vancomycin — Vancomycin 125mg orally four times per day for 12 days
  Arms: OF_UF Vancomycin; UF_OF Vancomycin
Drug: Placebo oral tablet — Placebo pills orally four times per day for 12 days
  Arms: OF_UF Placebo; UF_OF Placebo
Other: Overfeeding diet (OF) — Diet in which the calories are 150% of their weight maintaining energy requirements
Other: Underfeeding diet (UF) — Diet in which the calories are 50% of their weight maintaining energy requirements

SUMMARY:
We propose to study both stool and urine energy loss in 24 individuals on two experimental diets (50% increased and 50% reduced nutrient load relative to body size) in a random cross-over design. Following this over/underfeeding, volunteers will also be randomly assigned to a placebo versus oral antibiotic medication arm. This study will extend our previous findings by investigating whether 1) nutrient absorption changes upon similar increases/decreases in relative nutrient load and 2) whether manipulation of gut microbial communities with antibiotics alters nutrient absorption and 3) how these changes may affect glucose tolerance and fat storage.

DETAILED DESCRIPTION:
The prevalence of obesity has risen to epidemic proportions in the world, resulting from both excessive energy intake and low levels of energy expenditure. The effect of nutrient absorption on energy balance, that is, the relative amount of nutrients consumed vs. the amount excreted in stool, has been reported only in small studies in which energy waste in feces and urine between lean and obese individuals was not found to be different. New studies have shown that bacteria in the gut may play an important role in calorie absorption. We have recently shown that leaner individuals absorbed more calories when overfed compared to when they were given a diet with just enough calories to maintain their own weight. Our studies have also found that overfeeding also changes the kinds of bacteria found in the gut. In lean individuals, these changes in gut bacterial communities with overfeeding were associated with changes in how many calories were absorbed. Our results are similar to those seen in other studies in animals and humans that suggest a role for gut bacteria in weight gain and obesity. To try to better understand the role of gut bacteria in absorbing food, we propose to investigate 1) whether energy loss (as measured in stool and urine) changes following over- and underfeeding relative to body size and 2) whether changes in the gut bacteria, induced by an antibiotic medication, affect nutrient absorption and glucose tolerance. We plan to study 24 healthy non-smoking volunteers age 18 45 years old, not taking any medications (including medications for weight loss, antibiotics or probiotics) for the examination. All participants will be admitted to the Clinical Research Unit for 31 days. During their stay, subjects will be fed a weight maintaining diet for 3 days, followed by two experimental diets (150% and 50% of weight maintaining calories) in a random order. After this, volunteers will be randomly assigned to one of two groups: group 1 will take oral antibiotic medication; group 2 will receive pills that look the same but will not contain any active medication (placebos). Feces (stool) will be collected throughout the study. Additionally, twenty four-hour urine collections will take place each day of the experimental diet period and when stool is collected on the antibiotics. The energy content of these waste products as well as that of the diet (using duplicate plate analysis) will be measured by bomb calorimetry. Bacterial components in feces will be extracted by repeated fractional centrifugation to obtain bacterial mass and by using 16S rDNA-based oligonucleotide probes to obtain data on gut bacteria. Primary results will examine how many calories remain in stool during relative over- and underfeeding and whether changes in gut bacteria, induced by an antibiotic medication, affect nutrient absorption and glucose tolerance.

ELIGIBILITY:
* INCLUSION CRITERIA:

Free of acute and chronic diseases (especially GI disorders) as determined by medical history, physical examination and laboratory tests.

Individuals may be taking laxative drugs but they must be discontinued 3 or more weeks before admission.

Age 18-45 y (in order to minimize the affect of aging on nutrient absorption).

EXCLUSION CRITERIA:

Because it is unclear how chronic illnesses or substance abuse could affect nutrient absorption we will exclude volunteers with chronic diseases or current substance abuse. This is especially important because the limited number of study subjects in this study will make it hard to control for these confounders. We will therefore exclude subjects with a history or clinical manifestation of:

* Current smoking
* Type 2 diabetes (according to the World Health Organization diagnostic criteria)
* Endocrine disorders, such as Cushing s disease, pituitary disorders, and hypo- and hyperthyroidism
* HIV infection (self-report), due to effects on weight and body composition of HIV and medications used to treat HIV
* Active tuberculosis (self-report)
* Asthma on active daily treatment with medications
* Pulmonary disorders including physician diagnosed chronic obstructive pulmonary diseases and obstructive sleep apnea syndrome
* Cardiovascular diseases, including coronary heart disease, heart failure, arrhythmias, and peripheral artery disease
* Hypertension (according to the World Health Organization diagnostic criteria), treated or uncontrolled
* Gastrointestinal disease, including inflammatory bowel diseases (e.g. Crohn s disease and ulcerative colitis), malabsorption syndromes (e.g. celiac disease), gastric ulcer (active) and irritable bowel syndrome.
* Lactose intolerance
* Anemia (defined as hemoglobin < 11 mg/dl), leucopenia (defined as white blood cell count < 4,000/microL) or thrombocytopenia (defined as platelet count < 150,000/microL)
* Liver disease, including non-alcoholic fatty liver disease or current elevated liver enzymes over 1.5 times the normal range for AST, ALT or GGT or a history and physical exam that indicates a potential liver disease as describe by Giannini et al
* Evidence of chronic renal disease as defined by estimated glomerular filtration rate of < 60 ml/min or evidence of overt proteinuria on urine dipstick.
* Central nervous system disease, including previous history of cerebrovascular accidents, dementia, and neurodegenerative disorders
* Cancer requiring treatment in the past five years, except for non-melanoma skin cancers or cancers that have clearly been cured or in the opinion of the investigator carry an excellent prognosis
* Behavioral or psychiatric conditions that would be incompatible with a safe and successful participation in the study (such as major depression, schizophrenia and presence of psychotic symptoms)
* Eating disorders such as anorexia nervosa, bulimia or binge eating syndrome
* Taking weight loss drugs
* Weight change of more than 5% of total body weight in the 3 months before admission
* Use of any antibiotic or probiotic agents within 6 months prior to minimize the potential effects of these substances on the gut microbiota.
* Use of antacids (Proton pump inhibitors, H2 antagonists or aluminum/magnesium hydroxide) 3 months prior to the study assessed by self-report because a modified gastric pH might affect the gut microbiota as well
* Evidence of alcohol and/or drug abuse (more than 3 drinks per day and use of drugs, such as amphetamines, cocaine, heroin, or marijuana)

The following exclusion criteria are necessary because of the substances given or tests performed during the study

* Known allergies to vancomycin
* Known allergies to heparin or a history of heparin-induced thrombocytopenia
* Personal history or evidence of a bleeding disorder

All individuals will be fully informed of the aim, nature, and risks of the study prior to giving written informed consent. The study s informed consent will be obtained by a principal or associate investigator, research physician or physician assistant working in the clinical research unit.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2014-01-14; Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Krakoff, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Background] Yanovski SZ, Yanovski JA. Obesity. N Engl J Med. 2002 Feb 21;346(8):591-602. doi: 10.1056/NEJMra012586. No abstract available. PMID 11856799
- [Background] Weststrate JA, Dekker J, Stoel M, Begheijn L, Deurenberg P, Hautvast JG. Resting energy expenditure in women: impact of obesity and body-fat distribution. Metabolism. 1990 Jan;39(1):11-7. doi: 10.1016/0026-0495(90)90141-x. PMID 2294371
- [Background] Segal KR, Dunaif A. Resting metabolic rate and postprandial thermogenesis in polycystic ovarian syndrome. Int J Obes. 1990 Jul;14(7):559-67. PMID 2228390
- [Result] Basolo A, Hohenadel M, Ang QY, Piaggi P, Heinitz S, Walter M, Walter P, Parrington S, Trinidad DD, von Schwartzenberg RJ, Turnbaugh PJ, Krakoff J. Effects of underfeeding and oral vancomycin on gut microbiome and nutrient absorption in humans. Nat Med. 2020 Apr;26(4):589-598. doi: 10.1038/s41591-020-0801-z. Epub 2020 Mar 23. PMID 32235930
- [Derived] Basolo A, Parrington S, Ando T, Hollstein T, Piaggi P, Krakoff J. Procedures for Measuring Excreted and Ingested Calories to Assess Nutrient Absorption Using Bomb Calorimetry. Obesity (Silver Spring). 2020 Dec;28(12):2315-2322. doi: 10.1002/oby.22965. Epub 2020 Oct 7. PMID 33029899

RESULTS

PARTICIPANT FLOW:
Period: Phase 1: Crossover UF and OF
Arm/Group | OF_UF Vancomycin | OF_UF Placebo | UF_OF Vancomycin | UF_OF Placebo
Started | 9 | 7 | 4 | 7
Completed | 9 | 7 | 4 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Phase 2: Vancomycin and Placebo
Arm/Group | OF_UF Vancomycin | OF_UF Placebo | UF_OF Vancomycin | UF_OF Placebo
Started | 9 | 7 | 4 | 7
Completed | 8 | 7 | 4 | 6
Not Completed | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OF_UF Vancomycin | OF_UF Placebo | UF_OF Vancomycin | UF_OF Placebo | Total
Number analyzed (Participants) | 9 | 7 | 4 | 7 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (13.3) | 34.9 (7.2) | 29.7 (4.4) | 38.4 (3.6) | 35.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 3 | 10
  Male | 6 | 5 | 2 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 0 | 3
  Not Hispanic or Latino | 8 | 5 | 4 | 7 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 3 | 3 | 2 | 13
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 1 | 5
  White | 1 | 1 | 0 | 4 | 6
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Stool Calories During OF and UF
Description: Calculated as stool calories (kcal/day) x 100/ingested calories (kcal/day)
Time Frame: Days 5-7 and 11-13
Population: 4 subjects were excluded from the analysis because the delineation of the diet periods using two dye markers was not clear
Measure: Mean (Standard Deviation); unit: percentage of calorie intake
Groups:
- Overfeeding: Healthy volunteers assigned overfeeding diet
  Overfeeding diet (OF): Diet in which the calories are 150% of their weight maintaining energy requirements
- Underfeeding: Healthy volunteers assigned underfeeding diet
  Underfeeding diet (UF): Diet in which the calories are 50% of their weight maintaining energy requirements
Arm/Group | Overfeeding | Underfeeding
Number analyzed (Participants) | 23 | 23
percentage of calorie intake | 5.8 (1.9) | 8.9 (3.7)

2. Primary Outcome: Stool Calories During Vancomycin and Placebo
Description: Calculated as stool calories (kcal/day) x 100/ingested calories (kcal/day), vancomycin compared to placebo
Time Frame: Days 23-25
Population: Phase 2: Of the 27 participants enrolled, 2 participants dropped out and 1 had missing stool data
Measure: Mean (Standard Deviation); unit: percentage of calorie intake
Groups:
- Vancomycin: Healthy volunteers assigned overfeeding diet, underfeeding diet, and then vancomycin
  Vancomycin: Vancomycin 125mg orally four times per day for 12 days
  Overfeeding diet (OF): Diet in which the calories are 150% of their weight maintaining energy requirements
  Underfeeding diet (UF): Diet in which the calories are 50% of their weight maintaining energy requirements
- Placebo: Healthy volunteers assigned overfeeding diet, underfeeding diet, and then placebo
  Placebo oral tablet: Placebo pills orally four times per day for 12 days
  Overfeeding diet (OF): Diet in which the calories are 150% of their weight maintaining energy requirements
  Underfeeding diet (UF): Diet in which the calories are 50% of their weight maintaining energy requirements
Arm/Group | Vancomycin | Placebo
Number analyzed (Participants) | 11 | 13
percentage of calorie intake | 8.4 (1.9) | 5.6 (2.5)

3. Secondary Outcome: Urine Calories During OF and UF
Description: Calculated as urine calories (kcal/day) x 100/ingested calories (kcal/day)
Time Frame: Days 5-7 and 11-13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of calorie intake
Arm/Group | Overfeeding | Underfeeding
Number analyzed (Participants) | 23 | 23
percentage of calorie intake | 1.1 (0.2) | 2.3 (0.5)

4. Secondary Outcome: Urine Calories During Vancomycin and Placebo
Description: Calculated as urine calories (kcal/day) x 100/ingested calories (kcal/day), vancomycin compared to placebo
Time Frame: Days 23-25
Population: Phase 2: Of the 27 participants enrolled, 2 participants dropped out and 1 had missing stool data
Measure: Mean (Standard Deviation); unit: percentage of calorie intake
Arm/Group | Vancomycin | Placebo
Number analyzed (Participants) | 11 | 13
percentage of calorie intake | 1.3 (0.3) | 1.3 (0.2)

5. Secondary Outcome: Change in 2 Hour Glucose Tolerance From Day 16 to Day 28 During Vancomycin and Placebo
Description: A 75-g 2 hour oral glucose tolerance test (OGTT) was performed on days 16 and 28, before and after treatment with vancomycin or placebo.
Time Frame: Day 16 and day 28
Population: Phase 2: Of the 27 participants enrolled, 2 participants dropped out and 1 had a missing OGTT.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vancomycin | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL | 1.3 (16.8) | -1.9 (21.2)

6. Secondary Outcome: Overall Gut Microbial Colonization During OF and UF
Description: qPCR-based quantification of 16S rRNA gene copies per gram wet weight (log10)
Time Frame: Days 5-7 and 11-13
Population: Data were available during both diets for only 15 subjects
Measure: Median (Inter-Quartile Range); unit: log 10 copies per gram weight
Arm/Group | Overfeeding | Underfeeding
Number analyzed (Participants) | 15 | 15
log 10 copies per gram weight | 9.39 [9.21 to 9.98] | 9.73 [9.32 to 10.52]

7. Secondary Outcome: Overall Gut Microbial Colonization During Vancomycin and Placebo
Description: qPCR-based quantification of 16S rRNA gene copies per gram wet weight (log10)
Time Frame: Days 23-25
Population: Data were available for only 23 subjects
Measure: Median (Inter-Quartile Range); unit: log 10 copies per gram weight
Arm/Group | Vancomycin | Placebo
Number analyzed (Participants) | 11 | 12
log 10 copies per gram weight | 9.92 [9.41 to 10.14] | 9.42 [9.07 to 10.06]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 31 days
Description: All adverse events, including those observed by or reported to the research team, will be recorded. Serious unanticipated problems, Unanticipated Adverse Device Effects and serious protocol deviations, will be reported to the IRB and Clinical Director (CD) as soon as possible but not more than 7 days after the PI first learns of the event. Not serious unanticipated problems will be reported to the IRB and CD as soon as possible but not more than 14 days after the PI first learns of the event.
Groups:
- Overfeeding: Healthy volunteers assigned overfeeding diet (OF): Diet in which the calories are 150% of their weight maintaining energy requirements
- Underfeeding: Healthy volunteers assigned underfeeding diet (UF): Diet in which the calories are 50% of their weight maintaining energy requirements
- Vancomycin: Healthy volunteers assigned Vancomycin: Vancomycin 125mg orally four times per day for 12 days
- Placebo: Healthy volunteers assigned Placebo oral tablet: Placebo pills orally four times per day for 12 days
Arm/Group | Overfeeding | Underfeeding | Vancomycin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT02037295/Prot_SAP_000.pdf